CLINICAL TRIAL: NCT00995774
Title: Extension of the MIME Robotic System for Stroke Rehabilitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B4719-R
Record Dates: First submitted 2009-10-08; First posted 2009-10-15 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Stroke; Impaired Upper Extremity Function
Keywords: stroke; function; arm; hand; robotic; therapy; motor; movement; treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic then Conventional (Experimental): robotic arm therapy first, conventional therapy second
  Interventions: Device: robotic therapy; Other: conventional functional training
- Conventional then Robotic (Experimental): conventional therapy first, robotic therapy second
  Interventions: Device: robotic therapy; Other: conventional functional training

INTERVENTIONS:
Device: robotic therapy — 12 sessions of robot therapy for arm and hand function
  Arms: Robotic then Conventional
Other: conventional functional training — 12 sessions of conventional therapy for the arm and hand from a physical therapist
  Arms: Robotic then Conventional
Device: robotic therapy — 12 sessions of robot therapy for arm and hand function
  Arms: Conventional then Robotic
Other: conventional functional training — 12 sessions of conventional therapy for the arm and hand from a physical therapist
  Arms: Conventional then Robotic

SUMMARY:
The goal of this project is to develop and test a new robotic system to accommodate practice of tasks requiring reach, grasp and release of objects. Our previous work has shown that the MIME robot is safe and effective for improving reach in stroke subjects. But adequate control of hand movements is critical to a functional upper limb, and is often resistant to conventional therapeutic interventions. Many stroke survivors have residual ability to flex the fingers, but extension is often limited and impeded by increased passive stiffness in flexors, abnormal levels of increased tone in flexors and weakness in extensors. In a recent study, 38% of stroke survivors reported that impaired hand function was the most disabling motor impairment they faced.

DETAILED DESCRIPTION:
Research Design:

We hypothesize that: 1) Gains in proximal arm function (shoulder, elbow) immediately after robotic training will be greater than after dose-matched conventional therapy; 2) Unlike in previous studies, gains in hand function immediately after robotic training will be greater than after dose-matched conventional therapy.

Methodology:

In the first year of the study, we will develop a robotic system with the ability to assist hand movement. Since many stroke survivors in the subacute and chronic recovery stages have residual ability to flex the fingers but severely limited finger extension, we will build a hand exoskeleton that can apply precise extension forces to the digits of the hand. This exoskeleton will be integrated with the ARMin III arm exoskeleton so that tasks such as arm reach, grasp of an object and release of the object can be trained. In the last 2 years of the project, we will perform a pilot clinical trial comparing this new training paradigm to dose-matched conventional therapy in chronic stroke survivors. Outcome measures will be taken before training and immediately after training.

ELIGIBILITY:
Inclusion Criteria:

* An ischemic or hemorrhagic stroke more than 6 months prior to entry into the study;
* trace ability to move the wrist and fingers in extension;
* voluntary shoulder elevation to approximately 45 deg;
* be between the ages of 21 and 90.

Exclusion Criteria:

* Have cognitive deficits that could negatively affect their ability to complete protocols as evidenced by a score of 24 or less on the Folstein Mini - Mental State Examination (Bleeker, 1988);
* have excessive pain in any joint of the affected extremity that could limit ability to cooperate with the protocols;
* have an upper extremity injury or conditions prior to stroke that could limit participation;
* have severe hemispatial neglect.
* have a full score of 24 on the distal section of the Fugl-Myer test (FM) (Fugl-Meyer 1975); and
* have severe sensory loss.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S. Lum, PhD, Principal Investigator — VA Medical Center, DC
Locations (1):
- VA Medical Center, DC, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Brokaw EB, Nichols D, Holley RJ, Lum PS. Robotic therapy provides a stimulus for upper limb motor recovery after stroke that is complementary to and distinct from conventional therapy. Neurorehabil Neural Repair. 2014 May;28(4):367-76. doi: 10.1177/1545968313510974. Epub 2013 Dec 2. PMID 24297763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was through "word of mouth" with therapists at the outpatient clinics of the DC Veterans Affair Medical Center and the MedStar National Rehabilitation Hospital. Recruitment took place approximately between 9/2010 and 3/2012.
Pre-assignment Details: Fourteen individuals were recruited. One subject was excluded due to a prior orthopedic injury and another subject did not meet the Folstein Mini-Mental State Examination criterion. Two subjects completed the protocol up through the initial training period and the washout period, but did not return for the second therapy block.
Groups:
- Robotic Then Conventional: 12 hours of robotic arm therapy, followed by a 1 month washout period, followed by 12 hours of conventional arm therapy with a physical therapist
- Conventional Then Robotic: 12 hours of conventional arm therapy with a physical therapist, followed by a 1 month washout period, followed by 12 hours of robotic arm therapy
Period: Training Period 1
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0
Period: Training Period 2
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Started | 7 | 5
Completed | 5 | 5
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Then Conventional | Conventional Then Robotic | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.8) | 57.8 (16.3) | 57.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Test of Motor Function
Description: This scale assesses motor impairments at the shoulder, elbow, wrist and fingers (Fugl-Meyer 1975). Individual subscores are added to create a total score that ranges from 0 to 66 points. A score of 66 indicates no impairment.
Time Frame: before Training Period 1, after Training Period 1, before Training Period 2, after training Period 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Number analyzed (Participants) | 7 | 5
units on a scale
  Change from beginning to end of training period 1 | 1.9 (4.6) | .8 (2.9)
  Change from beginning to end of washout period | 1.3 (4.4) | .8 (3.9)
  Change from beginning to end of training period 2 | 1.6 (3.6) | 1.6 (2.3)

2. Secondary Outcome: Action Research Arm Test
Description: This scale is a standardized assessment of functional limitations in the upper extremity. Individual subscores are summed to create a total score that ranges from 0 to 57 points. A score of 57 indicates no functional limitations.
Time Frame: before Training Period 1, after Training Period 1, before Training Period 2, after training Period 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Number analyzed (Participants) | 7 | 5
units on a scale
  Change from beginning to end of training period 1 | 4.6 (3.5) | -.2 (1.1)
  Change from beginning to end of washout period | .4 (2.9) | 0 (1.6)
  Change from beginning to end of training period 2 | -2 (5.9) | 1.4 (3.0)

3. Secondary Outcome: A Motion Analysis Evaluation Will be Performed on Reach and Grasp Tasks. The Kinematics Will be Measured Using an Electromagnetic Tracker (Flock of Birds, Ascension Technology Corp., Burlington VT).
Time Frame: pre-treatment, post treatment
Population: Data initially collected but could not interpret results due to a lack of resources and incomplete data analysis. No further staff, tools, or information is available to report conclusions.
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Robotic Then Conventional | Conventional Then Robotic
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

LIMITATIONS AND CAVEATS:
The limited therapy hours could mask potential gains that would have been made with additional therapy. Due to the small sample size, these results need to be confirmed in a larger scale study using a parallel study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes